CLINICAL TRIAL: NCT00198497
Title: Phase III Safety and Efficacy Study of Vitrase (Ovine Hyaluronidase) for Ophthalmic Intravitreal Injection for Clearance of Severe Vitreous Hemorrhage
Brief Title: Safety and Efficacy Study of Vitrase for Clearance of Severe Vitreous Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIT-03-08961X
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Vitreous Hemorrhage; Diabetic Retinopathy
MeSH Terms: conditions — Vitreous Hemorrhage; Diabetic Retinopathy | interventions — Saline Solution; Chondroitinases and Chondroitin Lyases; Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrase (Experimental): Single Hyaluronidase ophthalmic intravitreal injection
  Interventions: Drug: Vitrase
- Placebo (Placebo Comparator): Single Saline solution intravitreal injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Other Names: Saline solution
  Arms: Placebo
Drug: Vitrase — Hyaluronidase 55 IU in saline solution
  Other Names: Hyaluronidase
  Arms: Vitrase
Drug: Vitrase — Hyaluronidase 75 IU in saline solution
  Other Names: Hyaluronidase
  Arms: Vitrase

SUMMARY:
The purpose of this study is to determine if intravitreal injection of Vitrase (ovine hyaluronidase) clears vitreous hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Severe vitreous hemorrhage that obscures visualization of the fundus on indirect ophthalmoscopy, that has been present >/= 1 month by history or exam
* BCVA is worse than 20/200 at time of screening

Exclusion Criteria:

* Corneal or lenticular abnormalities that preclude fundus observation
* Ongoing ocular infection, inflammation or history of herpetic corneal lesion
* Current or prior retinal detachment or retinal tears or breaks or intraocular tumor
* More than 1 severe vitreous hemorrhage within 6 months
* Previous vitrectomy for any reason
* Hemorrhage is exclusively pre-retinal, or old & organized
* Prior Vitrase for intravitreal injection in either eye
* No light perception in either eye at any time
* Known contraindications to study medication
* Sickle cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510
Dates: Start 1999-06; Primary Completion 2001-09 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Vitreous hemorrhage resolution | 3 months
  laser treatment of underlying cause of vitreous hemorrhage, or other surgical treatment, or documented evidence of macula & at least 180 degrees of vitreous base, that vitreous hemorrhage cause is resolved

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
Visual Acuity | 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (58):
- Australia (6):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - University of Sydney, Sydney, New South Wales
  - University of Sydney/Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
- Brazil (6):
  - Universidade Federal de Goiania, Goiânia, Goiás
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Universidade Federal do Parana, Curitiba, Paraná
  - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Universidade de Sao Paulo, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo, Escola Paulista e Medicina, São Paulo, São Paulo
- Hungary (6):
  - Semmelweiss University, Budapest
  - Central Army Hospital of the Hungarian Army, Budapest
  - Uzsoki Street Hospital of the Municipality of Capital, Budapest
  - Medical University of Debrecen, Debrecen
  - Medical University of Pecs, Pécs
  - University of Szeged, Albert Szent-Gyorgyi Medical University, Szeged
- Italy (3):
  - Universita degli Studi dell'Aguila, Coppito
  - Universita degli Studi di Firenze, Florence
  - Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia, Roma
- Netherlands (3):
  - University of Amsterdam, Amsterdam, AZ
  - University Hospital Rotterdam, Rotterdam, Gelderland
  - Academic Hospital Groningen, Groningen, GZ
- Poland (9):
  - Klinika Chorob Oczu, Bydgoszcz
  - Silesian School of Medicine, Bytom
  - Ophtalmology Clinic, Gdansk
  - Medical Academy, Lodz, Lodz
  - Ophthalmology Chair and Clinic, Lublin
  - Main Regional Hospital, Poznan
  - K. Marcinkowski University of Medical Sciences, Poznan
  - Medical Academy, Warsaw, Warsaw
  - Wroclaw University of Medicine, Wroclaw
- South Africa (9):
  - Addington Hospital, KwaKhangela, Durban
  - Joseph J. Krouse, MB, ChB, Alberton
  - James Acton, MB ChB, Bellville
  - Nasionale Hospital, Bloemfontein
  - Newlands Surgical Clinic, Cape Town
  - Groote Schuur Hospital, Cape Town
  - Kelvin N. Rivett, MB, ChB, East London
  - Louis P. Kruger, MB, ChB, Johannesburg
  - Pretoria Eye Institute, Pretoria
- Spain (4):
  - Instituto Oftalmologico de Alicante, Alicante
  - Hospital de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Fe, Valencia
- United Kingdom (12):
  - H. M. Stanley Hospital, St Asaph, Denbighshire
  - Sussex Eye Hospital, Brighton, East Sussex
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - East Surrey Hospital, Redhill, Surrey
  - Bristol Eye Hospital, Bristol
  - Hull Royal Infirmary, Hull
  - Royal Liverpool University Hospital, Liverpool
  - St. Thomas' Hospital, London
  - Kings College Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Oxford Eye Hospital, Oxford

REFERENCES:
- [Derived] Bhavsar AR, Grillone LR, McNamara TR, Gow JA, Hochberg AM, Pearson RK; Vitrase for Vitreous Hemorrhage Study Groups. Predicting response of vitreous hemorrhage after intravitreous injection of highly purified ovine hyaluronidase (Vitrase) in patients with diabetes. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4219-25. doi: 10.1167/iovs.07-1602. Epub 2008 Apr 25. PMID 18441312